CLINICAL TRIAL: NCT02423135
Title: Detection of Autologous DEHP (DiEthylHexyl Phthalate)-Free Blood Transfusion Using a Combination of Multiple Biomarkers in Different Matrices.
Brief Title: Detection of Autologous DEHP (DiEthylHexyl Phthalate)-Free Blood Transfusion in Anti-doping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Nicolas Leuenberger, Dr, PhD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Protocol 06/14; 12C14NL (Other Grant/Funding Number: World Anti-doping Agency)
Record Dates: First submitted 2014-10-13; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Transfusion Reaction
MeSH Terms: conditions — Transfusion Reaction | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blood bags without DEHP (Experimental): Intervention : Autologous blood transfusion
  Interventions: Biological: Autologous blood transfusion
- Blood bags with DEHP (Experimental): Intervention : Autologous blood transfusion
  Interventions: Biological: Autologous blood transfusion

INTERVENTIONS:
Biological: Autologous blood transfusion — Volunteers make a blood donation and after 36 days of storage this blood is re-infused in the same volunteers.

SUMMARY:
The aim of the proposed project is to perform a clinical study in which volunteers will receive autologous blood transfusions in DEHP-free blood bags.

ELIGIBILITY:
Inclusion Criteria:

* Have to fill the swiss blood donation formulary

Exclusion Criteria:

* Anemia
* Cardiovascular disease
* Neurologic disease
* Not performed a blood donation for 5 weeks ago the start of the study.
* Immunological disease

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Measurement of blood parameters profile, iron metabolism and genomic compounds | 1 month
  Blood profiling such as measurement of concentration of different blood cells and hemoglobin will be measured up to 15 days after blood-reinfusion. Concentration of free-iron, ferritin and hepcidin will be measured in plasma and serum up to 15 days after blood re-infusion.
  Concentration of circulating microRNAs will be measured in plasma also up to 15 days after blood re-infusion. All measures are compared.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Leuenberger, PhD, Principal Investigator — Swiss Laboratory for Doping Analyses
Locations (1):
- Swiss Laboratory for Doping Analyses, Épalinges, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Leuenberger N, Barras L, Nicoli R, Robinson N, Baume N, Lion N, Barelli S, Tissot JD, Saugy M. Hepcidin as a new biomarker for detecting autologous blood transfusion. Am J Hematol. 2016 May;91(5):467-72. doi: 10.1002/ajh.24313. Epub 2016 Apr 6. PMID 26822428